CLINICAL TRIAL: NCT07322185
Title: COMPARATIVE EFFECTS OF STECCO-FASCIAL MANIPULATION AND ROLFING STRUCTURAL INTEGRATION IN PATIENTS WITH PIRIFORMIS SYNDROME; A RANDOMIZED CLINICAL TRIAL
Brief Title: Comparative Effects of Stecco-fascial Manipulation and Rolfing Structural Integration in Patients With Piriformis Syndrome
Acronym: Piriformis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Danyal Ahmad (Other)
Responsible Party: Sponsor-Investigator, Danyal Ahmad, Head Of Department (HOD), University of Management and Technology Sialkot Pakistan
Organization: University of Management and Technology Sialkot Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: kuhs/dpt/umt-skt-026
Record Dates: First submitted 2025-12-22; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Piriformis Syndrome
Keywords: Stecco-fascial Manipulation; Rolfing Structural Integration; Piriformis Muscle Syndrome; Manual Lymphatic Drainage; Muscle Recruitment
MeSH Terms: conditions — Piriformis Muscle Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP A ( Stecco fascial Manipulation) (Experimental): GROUP A ( Stecco fascial Manipulation) containing 21 participants who will be given Stecco fascial Manipulation for 30 minutes along with the conventional physiotherapy.
  Interventions: Other: Experimental: GROUP A ( Stecco fascial Manipulation)
- GROUP B (Rolfing Structural Integration) (Experimental): GROUP B (Rolfing Structural Integration) containing 21 participants who were given Rolfing Structural Integration for 30 minutes along with the conventional physiotherapy.
  Interventions: Other: Experimental: GROUP B (Rolfing Structural Integration)

INTERVENTIONS:
Other: Experimental: GROUP A ( Stecco fascial Manipulation) — Stecco-fascial manipulation primary reduces pain, improves range of motion, restores normal muscle recruitment link in myofascial sequences, facilitates healing by improving microcirculation and lymphatic drainage.
  Arms: GROUP A ( Stecco fascial Manipulation)
Other: Experimental: GROUP B (Rolfing Structural Integration) — Rolfing structural integration improves posture, reduces pain, lengthens fascial planes and enhances the movement efficiency. This research will determine which approach is more effective in treating the patient with piriformis syndrome.
  Arms: GROUP B (Rolfing Structural Integration)

SUMMARY:
This study aims to compare the effectiveness of Stecco Fascial Manipulation and Rolfing Structural Integration in treating Piriformis syndrome, focusing on special outcomes like pain severity and functional outcomes.

comparison will be done to check the effectiveness of Stecco-fascial Manipulation and Rolfing Structural Integration on patients of both groups.

participants will:

1. get the treatment according to their respective groups
2. Both groups were given 4 sessions for 4 weeks.

DETAILED DESCRIPTION:
This study will be a randomized clinical trial with a sample size of 42 participants as calculated with g power tool with 5% of attrition added. Subjects will be obtained by non- probability convenient sampling based on the inclusion and exclusion criteria. Participants will be randomly assigned into two groups, 21 subjects in each group. The group A will receive the stecco fascial manipulation along with the conventional therapy while group B will receive the rolfing structural integration along with conventional therapy. The conventional physiotherapy protocol will include TENS applied with a Hot- pack for 10 minutes that will be followed by piriformis stretch.The data analysis will be done by IBM SPSS 26.0 version. To check the normality Shaprio- Wilk test will be used.

ELIGIBILITY:
Inclusion Criteria:

1. 25 to 45 age group.
2. For at least four weeks, there has been unilateral buttock discomfort, either with or without posterior thigh pain included buttock pain, pain that worsened when sitting.
3. Positive slump test and fair test decrease ranges of hip NPRS greater than

Exclusion Criteria:

1. Previous pelvic, ipsilateral hip, lumbar, or sacroiliac surgery that would have confused pain source.
2. Evidence of lumbar radiculopathy or another spinal condition that could be the origin of the symptoms (matching MRI/CT revealing nerve root compression or disc herniation). progressive neurologic disease or neuromuscular disease (e.g., peripheral neuropathy, myopathy, neuromuscular junction diseases)28.
3. During the research period, pregnancy or the planning of pregnancy (if interventions are employed) active pelvic or hip infection, malignancy, fracture, or systemic inflammation.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in Pain Intensity as Measured by the Numerical Pain Rating Rating Scale (NPRS) | 4 Weeks
  The Numerical Pain Rating Scale (NPRS) is a self-intensity on an 11-point scale, ranging from 0 (no pain) to 10 (worst possible pain). It is widely used in both clinical and research demonstrated strong reliability and validity in measuring Scale (NPRS) is a self-reported tool used to assess pain point scale, ranging from 0 (no pain) to 10 (worst possible pain). It is research settings for musculoskeletal conditions, strong reliability and validity in measuring both acute and chronic pain reported tool used to assess pain point scale, ranging from 0 (no pain) to 10 (worst possible pain). It is conditions, and it has both acute and chronic pain
Universal Goniometer | 4 Weeks
  A goniometer is an instrument used objective and reliable values that help evaluate mobility limitations i disorders such as piriformis syndrome used to measure joint range of motion (ROM). It provides objective and reliable values that help evaluate mobility limitations in musculoskeletal disorders such as piriformis syndrome.

SECONDARY OUTCOMES:
FAIR Test | 4 Weeks
  The FAIR (Flexion, Adduction, and Internal Rotation) test is a provocation test specifically designed for diagnosing piriformis syndrome. It reproduces symptoms by stretching the piriformis muscle, The FAIR (Flexion, Adduction, and Internal Rotation) test is a provocation test specifically designed for diagnosing piriformis syndrome. It reproduces symptoms by which may compress or irritate the sciatic nerve. The FAIR (Flexion, Adduction, and Internal Rotation) test is a provocation test specifically designed for diagnosing piriformis syndrome. It reproduces symptoms by sciatic nerve. This test has been validated as a reliable diagnostic too has been validated as a reliable diagnostic tool in piriformis-related case
Slump Test | 4 Weeks
  The Slump test is a neurodynamic examination used to assess neural tension, particularly performed by placing the patient in a seated slumped tension, particularly slumped position with controlled spinal and limb movements, helping to reproduce neurological symptoms The Slump test is a neurodynamic examination used to assess neural of the sciatic nerve. It is performed with controlled spinal and limb movements, helping to reproduce neurological symptoms associated with lumbosacral or piriformis with controlled spinal and limb movements, helping to reproduce neurological symptoms associated with lumbosacral or piriformis-related condition.

CONTACTS AND LOCATIONS:
Overall Officials: HAMZA ZAHID, MS OMPT, Principal Investigator — University of Management and Technology Sialkot Pakistan
Locations (3):
- Pakistan (3):
  - Raheem Surgical Hospital Sambrial, Sambrial, Punjab Province
  - Bethania Hospital Sialkot, Sialkot, Punjab Province
  - University of Management and technology Sialkot Campus, Sialkot, Punjab Province

IPD SHARING:
Plan to Share IPD: Undecided